CLINICAL TRIAL: NCT00564642
Title: Investigation of the Effect of N Acetylcysteine Against Anti-Tuberculosis Drugs Induced Liver Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Institute of Tuberculosis and Lung Disease, Iran (Other Government)
Responsible Party: Dr. Baniasadi, National Research Institute of Tuberculosis and Lung Disease
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5344-21-07-86
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Hepatitis; Tuberculosis
MeSH Terms: conditions — Hepatitis; Tuberculosis | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: N Acetylcysteine — 1200 mg, BD, 2weeks
  Other Names: ACC

SUMMARY:
Tuberculosis is one of the major health problems in developing countries. Isoniazid, rifampin and pyrazinamide, the first line drugs used for tuberculosis chemotherapy, are associated with hepatotoxicity. The rate of hepatotoxicity has been reported to be much higher in developing countries compared to that in advanced countries with a similar dose schedule. Oxidative stress has proposed as one of the mechanisms responsible for anti-tuberculosis drugs induced hepatic injury. The oxidative stress is closely associated with decrease of glutathione levels. In the present study N acetylcysteine, a precursor of glutathione, was investigated for hepatoprotective effect against anti-tuberculosis drugs induced liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Two sputum specimens positives for tubercle bacilli on direct smear microscopy
* No previous anti-TB chemotherapy higher than two weeks
* Aged 60 years and over
* Agreement to participate in the study

Exclusion Criteria:

* Alcohol consumption
* Viral disease (Hepatitis,...)
* Abnormal pretreatment LFT level
* Chronic disease (liver and kidney disease, asthma,...)
* Additional hepatotoxic drug use
* HIV positive
* Liver TB
* Patient in a moribund state
* Hemoptysis

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Hepatotoxicity | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Baniasadi, PhD, Principal Investigator — National Research Institute of Tuberculosis and Lung Disease (NRITLD)-Shaheed Beheshti University of Medical Sciences
Locations (1):
- National Research Institute of Tuberculosis and Lung Disease (NRITLD), Tehran, Iran